CLINICAL TRIAL: NCT06757335
Title: A Multicenter, Open, Dose Escalation/dose Escalation, and Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral HP568 Tablets Alone and in Combination with Palbociclib in Patients with ER+/HER2 Advanced Breast Cancer
Brief Title: A Phase I/II Trial to Evaluate Oral HP568 Tablets in Patients with ER+/HER2 Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP568-101
Record Dates: First submitted 2024-11-07; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HP568 (Experimental): In the I/II stage: HP568 administered QD or BID for 28 day cycles.
  Interventions: Drug: HP568
- HP568 and palbociclib (Experimental): In the III stage: Daily oral dosages of HP568 for 28 days in combination with palbociclib for 21 days.
  Interventions: Drug: HP568 in combination with palbociclib

INTERVENTIONS:
Drug: HP568 — In the I/II stage: HP568 administered QD or BID for 28 day cycles.
  Arms: HP568
Drug: HP568 in combination with palbociclib — In the III stage: Daily oral dosages of HP568 for 28 days in combination with palbociclib for 21 days.
  Arms: HP568 and palbociclib

SUMMARY:
This is a Phase 1/2 dose escalation and cohort expansion study and will assess the safety, tolerability and preliminary efficacy of HP568 alone and in combination with palbociclib in patients with ER+/HER2- locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years old (inclusive of both ends) at the time of signing the informed consent form.
2. Patients with locally advanced inoperable or recurrent or metastatic breast cancer ER+/HER2- advanced breast cancer is confirmed by histopathology have confirmed that the primary and/or metastatic lesion.
3. Previously received at least 1-line endocrine therapy (endocrine therapy duration ≥ 6 months) and ≤ 2-line chemotherapy (≤ 2-line chemotherapy limited to dose escalation stage) for the recurrence or metastasis stage of the disease. The third stage : Inclusion of patients who have not received prior treatment but are suitable for CDK4/6i therapy.
4. Disease progression confirmed by imaging occurs during or after the last systemic anti-tumor treatment before the first medication.

Exclusion Criteria:

1. Known or suspected allergy to any ingredient of HP568 formulation, and allergy to any ingredient of palbociclib (only applicable to stage III).
2. Within 42 days prior to the first administration, Fluvistran was used; Other endocrine therapies such as tamoxifen, toremifene, letrozole, anastrozole, and exemestane were used within 14 days prior to the first administration.
3. Previously received other ER-ROTAC drugs such as ARV-471.
4. Within 6 weeks before the first administration of HP568 in this study, nitrosoureas or mitomycin were used; Received any anti-tumor treatment, including immunotherapy, chemotherapy, radiotherapy, or targeted therapy, within 28 days prior to the first administration (or of the drug's 5 half lives,take the shorter one).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Stage I: the incidence of TEAE of HP568 | From the first administration dose to 30 calendar days after the last administration dose
  the percentage of patients with treatment-emergent Adverse events(TEAE), TEAE will be evaluated using CTCAE 5.0 standards.
Stage I: Incidence of dose limiting toxicity DLT, maximum tolerated dose MTD (if possible). | 28 days
  First cycle dose-limiting toxicities and determination of a maximum tolerated dose (MTD) if applicable among the doses evaluated
Stage III: Evaluate safety during the dose escalation phase of combination therapy | From the first administration dose to 30 calendar days after the last administration dose
  Adverse events will be evaluated using the CTCAE5.0 standard, and safety features will be based on the assessment of adverse events, including TEAE, laboratory indicators (blood routine, blood biochemistry, coagulation routine, blood lipids, urine routine), vital sign measurements (blood pressure, pulse, respiratory rate, and body temperature), physical examination, and 12 lead electrocardiogram.
Stage III: Evaluate tolerance during the dose escalation phase of combination therapy | 28 days
  First cycle dose-limiting toxicities and determination of a maximum tolerated dose (MTD) if applicable among the doses evaluated
Stage III: Evaluate the 24 week clinical benefit rate (CBR) during the dose escalation phase of combination therapy | Until all patients have completed 24 weeks administration
  According to RECIST 1.1 criteria, the proportion of subjects who achieve confirmed CR (complete response) and/or confirmed PR (partial response) within 24 weeks plus at least 24 weeks of SD (stable disease).
Stage II: 24 week clinical benefit rate (CBR) | Until all patients have completed 24 weeks administration
  According to RECIST 1.1 criteria, the proportion of subjects who achieve confirmed CR (complete response) and/or confirmed PR (partial response) within 24 weeks plus at least 24 weeks of SD (stable disease).

SECONDARY OUTCOMES:
Stage I-III: Objective response rate (ORR) | Until all patients have completed study（approximately 2 years）
  According to RECIST 1.1 criteria, the proportion of subjects who achieve CR (complete response)+PR (partial response).
Stage I/III: 24 week clinical benefit rate (CBR) | Until all patients have completed 24 weeks administration
  According to RECIST 1.1 criteria, the proportion of subjects who achieve confirmed complete response (CR) and/or confirmed partial response (PR) within 24 weeks plus at least 24 weeks of stable disease (SD).
Stage I-III: Disease Control Rate (DCR) | Until all patients have completed study（approximately 2 years）
  The proportion of subjects who achieve response and disease stability (i.e. CR+PR+SD) after treatment.
Stage I-III: Progression free survival (PFS) | Until all patients have completed study（approximately 2 years）
  from the start of treatment until tumor progression or death from any cause, which comes first.
Stage I-III: Duration of response(DOR) | Until all patients have completed study（approximately 2 years）
  the time from the first onset of response (CR or PR) to disease progression
Stage I-III: Time to Response (TTR) | Until all patients have completed study（approximately 2 years）
  The time from the start of treatment to the first recorded achievement of response (CR or PR).
Stage I-II：Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC) | on the first day of cycle 1 and cycle 2（each cycle is 28 days）
  Concentration-time curve (AUC) for single and multiple dose of HP568 will be assessed after a single dose and after multiple doses.
Stage I-II：Assessment of pharmacokinetic parameter maximum concentration (Cmax) | on the first day of cycle 1 and cycle 2（each cycle is 28 days）
  Maximum concentration (Cmax) for single and multiple dose of HP568 will be assessed after a single dose and after multiple doses.
Stage I-II: Assessment of pharmacokinetic parameter minimum concentration (Cmin). | on the first day of cycle 1 and cycle 2 (each cycle is 28 days)
  minimum concentration (Cmin) for single and multiple dose of HP568 will be assessed after a single dose and after multiple doses.
Stage I-II：Assessment of pharmacokinetic parameter time to maximum concentration (Tmax) | on the first day of cycle 1 and cycle 2 (each cycle is 28 days)
  Time to maximum concentration (Tmax) for HP568 will be assessed after a single dose and after multiple doses.
Stage III：Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC) | on the Day 1 and Day 21 of cycle 1 (each cycle is 28 days)
  Concentration-time curve (AUC) of HP568 and palbociclib will be assessed after single and multiple doses.
Stage III: Assessment of pharmacokinetic parameter maximum concentration (Cmax) | on the Day 1 and Day 21 of cycle 1 (each cycle is 28 days)
  maximum concentration (Cmax) of HP568 and palbociclib will be assessed after a single dose and after multiple doses
Stage III: Assessment of pharmacokinetic parameter minimum concentration (Cmin) | on the Day 1 and Day 21 of cycle 1 (each cycle is 28 days)
  Minimum concentration (Cmin) of HP568 and palbociclib will be assessed after a single dose and after multiple doses.
Stage III: Assessment of pharmacokinetic parameter time to maximum concentration (Tmax) | on the Day 1 and Day 21 of cycle 1 (each cycle is 28 days)
  Time to maximum concentration (Tmax) of HP568 and palbociclib will be assessed after a single dose and after multiple doses.

IPD SHARING:
Plan to Share IPD: No